CLINICAL TRIAL: NCT05622812
Title: A Randomized, Evaluator-blinded, Parallel Group, no Treatment Controlled, Multicenter Study to Evaluate Effectiveness and Safety of Restylane Lyft Lidocaine for Jawline Definition
Brief Title: Effectiveness and Safety of Restylane Lyft Lidocaine for Jawline Definition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05DF2209
Record Dates: First submitted 2022-11-07; First posted 2022-11-21 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Jawline Definition

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, evaluator-blinded, no treatment controlled, parallel group, multicenter phase IV study to evaluate effectiveness and safety of Restylane Lyft Lidocaine for jawline definition.
  A parallel study: two or more groups of participants receive different interventions. Trial participants are assigned to one of the treatment arms at the beginning of the trial and remain in that trial arm throughout the length of the trial. A randomized group is usually assigned.
Who Masked: Outcomes Assessor
Masking Description: Investigator blinding will be accomplished by having a Treating Investigator administer the treatments and having a Blinded Evaluator, to whom randomization and treatment are concealed, conduct blinded assessments.
  Investigator blinding will be accomplished by having a Treating Investigator administer the treatments and having a Blinded Evaluator, to whom randomization and treatment are concealed, conduct blinded assessments. Safety assessments will be performed by non-blinded personnel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Initial Restylane Lyft Lidocaine injection and one optional touch-up treatment at 1 month after treatment
  Interventions: Device: Restylane Lyft Lidocaine
- No-treatment control group (No Intervention): Optional treatment will be administered at 12 months

INTERVENTIONS:
Device: Restylane Lyft Lidocaine — Treatment for Jawline definition
  Arms: Treatment group

SUMMARY:
This study is designed to evaluate effectiveness and safety of Restylane Lyft Lidocaine for Jawline definition

DETAILED DESCRIPTION:
A randomized, evaluator-blinded, parallel group, no treatment controlled, multicenter study to evaluate effectiveness and safety of Restylane Lyft Lidocaine for Jawline definition in Canada

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults willing to comply with the requirements of the study and providing a signed written informed consent
* Consent the use of facial images for marketing purposes and educational material
* Subject with moderate to very severe (Grade 2 to 4) on the GJS
* Subject is willing to abstain from any other facial, submental, and/or neck aesthetic procedure(s) or implant
* Female of childbearing potential with a negative urine pregnancy test before treatment

Exclusion Criteria:

* Subjects presenting with known/previous allergy or hypersensitivity to hyaluronic acid (HA) filler, lidocaine or other amide-type local anesthetics
* Subjects presenting with known/previous allergy or hypersensitivity to streptococcal proteins
* Subject with bleeding disorders or taking thrombolytics or anticoagulants
* Prior surgical procedure in the treatment area
* History of other facial treatment/procedure in the previous 6 months HA in or near the intended treatment site
* Presence of any disease or lesions near or on the area to be treated
* Presence of any condition, in the opinion of the Treating Investigator, makes the subject unable to complete the study per protocol
* Women who are pregnant or breast feeding, or women of childbearing potential who are not practicing adequate contraception or planning to become pregnant during the study period
* Study site personnel, close relatives of the study site personnel, employees, or close relatives of employees at the Sponsor Company
* Participation in any other interventional clinical study within 30 days before treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2024-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Galderma R&D
Locations (8):
- Canada (8):
  - Galderma Research Site, Vancouver, British Columbia
  - Galderma Research Site, Burlington, Ontario
  - Galderma Research Site, London, Ontario
  - Galderma Research Site, Oakville, Ontario
  - Galderma Research Site, Toronto, Ontario
  - Galderma Research Site, Windsor, Ontario
  - Galderma Research Site, Woodbridge, Ontario
  - Galderma Research Site, Westmount, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 9 sites in Canada from 16 February 2023 to 14 June 2024.
Pre-assignment Details: A total of 150 participants were screened, of which 10 were screen failures. A total of 140 participants were enrolled and randomized in the study.
Groups:
- Restylane Lyft Lidocaine: Participants received Restylane Lyft Lidocaine injection at Day 1 and one optional touch-up treatment at 1 month after treatment.
- No-treatment Control Group: Participants remained untreated and were offered optional treatment at 12 months from Baseline (Day 1).
Period: Overall Study
Arm/Group | Restylane Lyft Lidocaine | No-treatment Control Group
Started | 105 | 35
Completed | 102 | 30
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on the intent-to-treat (ITT) population. The ITT population included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Restylane Lyft Lidocaine | No-treatment Control Group | Total
Number analyzed (Participants) | 105 | 35 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (10.82) | 53.2 (11.13) | 54.7 (10.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 32 | 130
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 103 | 32 | 135
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 0 | 3
  White | 94 | 32 | 126
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders Having At Least a 1-Grade Improvement From Baseline on Both Jawlines Concurrently Based on Galderma Jawline Scale (GJS) at Month 3 as Assessed by Blinded Evaluator
Description: The GJS is a validated 5-point scale (ranges 0-4) for assessment of the jawline. Each score in the GJS is represented by photographic images of the scale, where 0 = none to minimal, 1 = mild, 2 = moderate, 3 = severe and 4 = very severe volume deficiency posterior to the jowl along the jawline. The Blinded Evaluator performed live assessment of the participant's left and right jawline separately. Here, a higher score indicated more volume deficiency in the treatment area. A responder was defined as participants having at least a 1-grade improvement from baseline on both jawlines concurrently.
Time Frame: Baseline, Month 3
Population: Analysis was performed on ITT population. The ITT population included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Restylane Lyft Lidocaine | No-treatment Control Group
Number analyzed (Participants) | 105 | 35
percentage of responders | 67.6 [57.8 to 76.4] | 28.6 [14.6 to 46.3]
Statistical Analysis 1: Comparison: Restylane Lyft Lidocaine vs No-treatment Control Group; Test type: Superiority; p < 0.001, Fisher's Exact Test. — Two-sided p-value calculated using Fisher's Exact Test. The threshold of significance at <0.05; Treatment difference = 39.0, 95% CI 2-sided [21.6 to 56.5] — Difference confidence interval calculated using normal approximation

2. Secondary Outcome: Percentage of Responders Having at Least a 1-Grade Improvement From Baseline on Both Jawlines Concurrently Based on GJS at Month 6, 9 and 12 as Assessed by Blinded Evaluator
Description: The GJS is a validated 5-point scale for assessment of the jawline. Each score in the GJS is represented by photographic images of the scale, where 0 = none to minimal, 1 = mild, 2 = moderate, 3 = severe and 4 = very severe volume deficiency posterior to the jowl along the jawline. Here, higher score indicated more volume deficiency in the treatment area. A responder was defined as participants having at least a 1-grade improvement from baseline on both jawlines concurrently.
Time Frame: Baseline, Months 6, 9 and 12
Population: Analysis was performed on ITT population. The ITT population included all participants who were randomized. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Restylane Lyft Lidocaine | No-treatment Control Group
Number analyzed (Participants) | 102 | 32
percentage of responders
  Month 6: number analyzed (Participants) | 98 | 32
  Month 6 | 62.2 [51.9 to 71.8] | 21.9 [9.3 to 40.0]
  Month 9: number analyzed (Participants) | 102 | 31
  Month 9 | 57.8 [47.7 to 67.6] | 16.1 [5.5 to 33.7]
  Month 12: number analyzed (Participants) | 101 | 31
  Month 12 | 49.5 [39.4 to 59.6] | 19.4 [7.5 to 37.5]
Statistical Analysis 1: Comparison: Restylane Lyft Lidocaine vs No-treatment Control Group; Month 6; Test type: Superiority; p < 0.001, Fisher's Exact Test. — Two-sided p-value calculated using Fisher's Exact Test. The threshold of significance at <0.05; Treatment difference = 40.4, 95% CI 2-sided [23.1 to 57.6] — Difference confidence interval calculated using normal approximation
Statistical Analysis 2: Comparison: Restylane Lyft Lidocaine vs No-treatment Control Group; Month 9; Test type: Superiority; p < 0.001, Fisher's Exact Test. — Two-sided p-value calculated using Fisher's Exact Test. The threshold of significance at <0.05; Treatment difference = 41.7, 95% CI 2-sided [25.6 to 57.8] — Difference confidence interval calculated using normal approximation
Statistical Analysis 3: Comparison: Restylane Lyft Lidocaine vs No-treatment Control Group; Month 12; Test type: Superiority; p = 0.003, Fisher's Exact Test. — Two-sided p-value calculated using Fisher's Exact Test. The threshold of significance at <0.05; Treatment difference = 30.2, 95% CI 2-sided [13.2 to 47.1] — Difference confidence interval calculated using normal approximation

3. Secondary Outcome: Percentage of Participants Having at Least "Improved" on the Global Aesthetic Improvement Scale (GAIS) on Both Jawlines Concurrently, as Assessed Live by the Treating Investigator at Months 3, 6, 9 and 12
Description: The 7-graded GAIS was used to live assess the aesthetic improvement of the jawline, that is, an improvement from baseline appearance before the first treatment by the Treating Investigator and the Participant, independently of each other. The participant responded to the question: "How would you describe the aesthetic improvement of the treatment area today compared to the photograph taken before treatment?" by using the categorical scale: Very Much Improved, Much Improved, Improved, No Change, Worse, Much Worse and Very Much Worse. Percentage of participants having at least "Improved" on the GAIS as assessed live by the Treating Investigator was reported here.
Time Frame: Baseline, Months 3, 6, 9 and 12
Population: Analysis was performed on the ITT population. The ITT population included all randomized participants. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Restylane Lyft Lidocaine | No-treatment Control Group
Number analyzed (Participants) | 102 | 33
percentage of participants
  Month 3 | 99.0 [94.7 to 100.0] | 0.0 [0.0 to 10.6]
  Month 6: number analyzed (Participants) | 99 | 32
  Month 6 | 97.0 [91.4 to 99.4] | 9.4 [2.0 to 25.0]
  Month 9: number analyzed (Participants) | 102 | 31
  Month 9 | 90.2 [82.7 to 95.2] | 9.7 [2.0 to 25.8]
  Month 12: number analyzed (Participants) | 102 | 30
  Month 12 | 80.4 [71.4 to 87.6] | 6.7 [0.8 to 22.1]
Statistical Analysis 1: Comparison: Restylane Lyft Lidocaine vs No-treatment Control Group; Month 3; Test type: Superiority; p < 0.001, Fisher's Exact Test. — Two-sided p-value calculated using Fisher's Exact Test. The threshold of significance at <0.05; Treatment difference = 99.0, 95% CI 2-sided [97.1 to 100.0] — Difference confidence interval calculated using normal approximation
Statistical Analysis 2: Comparison: Restylane Lyft Lidocaine vs No-treatment Control Group; Month 6; Test type: Superiority; p < 0.001, Fisher's Exact Test. — Two-sided p-value calculated using Fisher's Exact Test. The threshold of significance at <0.05; Treatment difference = 87.6, 95% CI 2-sided [76.9 to 98.2] — Difference confidence interval calculated using normal approximation
Statistical Analysis 3: Comparison: Restylane Lyft Lidocaine vs No-treatment Control Group; Month 9; Test type: Superiority; p < 0.001, Fisher's Exact Test. — Two-sided p-value calculated using Fisher's Exact Test. The threshold of significance at <0.05; Treatment difference = 80.5, 95% CI 2-sided [68.6 to 92.4] — Difference confidence interval calculated using normal approximation
Statistical Analysis 4: Comparison: Restylane Lyft Lidocaine vs No-treatment Control Group; Month 12; Test type: Superiority; p < 0.001, Fisher's Exact Test. — Two-sided p-value calculated using Fisher's Exact Test. The threshold of significance at <0.05; Treatment difference = 73.7, 95% CI 2-sided [61.9 to 85.5] — Difference confidence interval calculated using normal approximation

4. Secondary Outcome: Percentage of Participants Having at Least "Improved" on the GAIS on Both Jawlines Concurrently, as Assessed Live by the Participant at Months 3, 6, 9 and 12
Description: The 7-graded GAIS was used to live assess the aesthetic improvement of the jawline, that is, an improvement from baseline appearance before the first treatment by the Treating Investigator and the Participant, independently of each other. The participant responded to the question: "How would you describe the aesthetic improvement of the treatment area today compared to the photograph taken before treatment?" by using the categorical scale: Very Much Improved, Much Improved, Improved, No Change, Worse, Much Worse and Very Much Worse. Percentage of participants having at least "Improved" on the GAIS as assessed live by the participant was reported here.
Time Frame: Baseline, Months 3, 6, 9 and 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Restylane Lyft Lidocaine | No-treatment Control Group
Number analyzed (Participants) | 102 | 33
percentage of participants
  Month 3 | 93.1 [86.4 to 97.2] | 0.0 [0.0 to 10.6]
  Month 6: number analyzed (Participants) | 99 | 32
  Month 6 | 87.9 [79.8 to 93.6] | 0.0 [0.0 to 10.9]
  Month 9: number analyzed (Participants) | 102 | 31
  Month 9 | 80.4 [71.4 to 87.6] | 0.0 [0.0 to 11.2]
  Month 12: number analyzed (Participants) | 102 | 31
  Month 12 | 71.6 [61.8 to 80.1] | 0.0 [0.0 to 11.2]
Statistical Analysis 1: Comparison: Restylane Lyft Lidocaine vs No-treatment Control Group; Month 3; Test type: Superiority; p < 0.001, Fisher's Exact Test. — Two-sided p-value calculated using Fisher's Exact Test. The threshold of significance at <0.05; Treatment difference = 93.1, 95% CI 2-sided [88.2 to 98.0] — Difference confidence interval calculated using normal approximation
Statistical Analysis 2: Comparison: Restylane Lyft Lidocaine vs No-treatment Control Group; Month 6; Test type: Superiority; p < 0.001, Fisher's Exact Test. — Two-sided p-value calculated using Fisher's Exact Test. The threshold of significance at <0.05; Treatment difference = 87.9, 95% CI 2-sided [81.4 to 94.3] — Difference confidence interval calculated using normal approximation
Statistical Analysis 3: Comparison: Restylane Lyft Lidocaine vs No-treatment Control Group; Test type: Superiority; p < 0.001, Fisher's Exact Test. — Two-sided p-value calculated using Fisher's Exact Test. The threshold of significance at <0.05; Treatment difference = 80.4, 95% CI 2-sided [72.7 to 88.1] — Difference confidence interval calculated using normal approximation
Statistical Analysis 4: Comparison: Restylane Lyft Lidocaine vs No-treatment Control Group; Month 12; Test type: Superiority; p < 0.001, Fisher's Exact Test. — Two-sided p-value calculated using Fisher's Exact Test. The threshold of significance at <0.05; Treatment difference = 71.6, 95% CI 2-sided [62.8 to 80.3] — Difference confidence interval calculated using normal approximation

ADVERSE EVENTS:
Time Frame: From Baseline up to 12 months after last treatment
Description: The Safety population included all participants who were treated with Restylane Lyft Lidocaine or were randomized to the No Treatment group at Baseline.
Arm/Group | Restylane Lyft Lidocaine | No-treatment Control Group
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/35
Serious Adverse Events (participants affected / at risk) | 2/105 | 1/35
Other Adverse Events (participants affected / at risk) | 39/105 | 12/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Restylane Lyft Lidocaine (N=105) | No-treatment Control Group (N=35)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Restylane Lyft Lidocaine (N=105) | No-treatment Control Group (N=35)
Injection site nodule (General disorders) | 5 | 0
Injection site discomfort (General disorders) | 1 | 0
Injection site pain (General disorders) | 2 | 0
Injection site swelling (General disorders) | 1 | 0
Injection site cyst (General disorders) | 1 | 0
Injection site inflammation (General disorders) | 1 | 0
Injection site mass (General disorders) | 1 | 0
Injection site papule (General disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
COVID-19 (Infections and infestations) | 5 | 2
Nasopharyngitis (Infections and infestations) | 5 | 3
Influenza (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Labyrinthitis (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 2 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 0
Migraine (Nervous system disorders) | 1 | 1
Device breakage (Product Issues) | 1 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 | 0
Urogenital prolapse (Reproductive system and breast disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Actinic cheilitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Postmenopause (Social circumstances) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT05622812/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT05622812/SAP_001.pdf